CLINICAL TRIAL: NCT03880331
Title: Prospective Randomized Clinical Trial Comparing Outcomes of Secondary Intention Wound Care Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey Tiger, Principal Investigator, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20193001
Record Dates: First submitted 2019-02-12; First posted 2019-03-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Wound Surgical; Wound Heal
Keywords: Secondary intention; Wound care methods
MeSH Terms: conditions — Surgical Wound | interventions — Debridement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded investigator will assess photographs of completely healed wounds
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive Debridement (Active Comparator): Aggressive and frequent debridement of fibrin and crust from the wound base down to pinpoint bleeding, both by the patient as part of daily wound care at home, and also by the clinician (either physician or experienced dermatologic surgery nurse) during follow-up visits. Silver nitrate will be used to treat excessive granulation tissue only if the granulation tissue is higher than the level of surrounding skin. Patients will return weekly until healed. Patients will be provided with detailed instructions and guidelines to help determine whether healing has taken place.
  Interventions: Procedure: Debridement
- Minimal Debridement (Active Comparator): No debridement of fibrin by the patient or the clinician. Exceptions include debridement of dried crust or eschar. Silver nitrate will be used to treat excessive granulation tissue only if the granulation tissue is higher than the level of surrounding skin. Patients will return every two weeks until healed. In between visits at weekly intervals, the patient will be contacted by phone to determine if healing has occurred in between clinic visits11. Patients will be provided with detailed instructions and guidelines to help determine whether healing has taken place.
  Interventions: Procedure: Debridement

INTERVENTIONS:
Procedure: Debridement — Aggressive vs Minimal Debridement

SUMMARY:
This is a randomized controlled trial which is designed to determine whether aggressive and frequent debridement of an acute post-surgical wound shortens healing time.

DETAILED DESCRIPTION:
Secondary intention is an established method of allowing post-surgical defects to heal. Previous studies have shown a positive association between the frequency of debridement and healing rates in chronic wounds. However, the effect of debridement on acute, post-surgical wounds is not well-described in the literature.

This randomized controlled trial is designed to determine whether aggressive and frequent debridement of an acute post-surgical wound shortens healing time.

ELIGIBILITY:
Inclusion Criteria:

1. Dermatology patients at Lahey Clinic:
2. who have undergone Mohs surgery or excision
3. who are older than 18 years
4. who are able to give consent
5. who had postoperative defects allowed to heal by secondary intention on the a) head and neck, b) trunk and upper extremities, c) lower extremities
6. who are willing and able to return to clinic in Peabody, MA, for all wound care visits

Exclusion Criteria:

1. Unable to consent (due to language barrier or mental status)
2. Unable to perform daily wound care
3. Unwilling or unable to return for follow-up
4. Have baseline venous stasis or pitting edema of the affected limb
5. Wear compression stockings or require use of a compressive bandage (such as an Unna Boot) at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Time to healing | 0-16 weeks
  Time to complete healing as determined by one of the study investigators

SECONDARY OUTCOMES:
Patient satisfaction with scar: Patient Scar Assessment Questionnaire (PSAQ) | 0-16 weeks. NOTE: The PSAQ will be completed by the patient once their wound is determined to be completely healed by the study investigators; usually between 6-8 weeks.
  As assessed by the Patient Scar Assessment Questionnaire (PSAQ), a validated questionnaire used standardly in Dermatology for assessing patient-based outcome measures of scarring. It consists of 5 subscales: appearance, symptoms consciousness, satisfaction with appearance and satisfaction with symptoms. Each subscale consists of a set of items with 4-point categorical responses, scoring 1 to 4 points (with 1 point assigned to the most favorable category and 4 assigned to the least favorable). It has been demonstrated to be a reliable and valid measure of patients' perception of scarring. See reference #12 in reference list for more information.
Cosmetic Appearance | 0-16 weeks. NOTE: A photograph of the the patient's final healed wound will be evaluated by a blinded investigator after the wound is determined to be completely healed by the study investigators; usually between 6-8 weeks
  As assessed by the Visual Analog Scale, a validated image-based scale, that uses photographs for evaluation in 5 dimensions (pigmentation, vascularity, acceptability, observer comfort, and contour). "Observer comfort" measures the observer's "comfort level" when viewing the wound. The benefit of using this scale for the purposes of the study is because it is a photograph-based scale which can be evaluated later by a blinded physician rather than in the clinic at the time of the visit. The observer places a mark along a continuous line that measures 10cm long, and then that is measured from left to right and a corresponding score is given corresponding to that length (between 0 and 10). The individual scores are tallied to obtain a single overall score ranging from "poor" to "excellent." See reference #13 in reference list for more information.
Number of required debridements | 0-16 weeks
  Number of required debridements over the course of healing
Number of treatment failures | Through study completion, an average of 6-8 weeks
  Number of wounds that do not heal by 16 weeks
Complications | 0-16 weeks
  Including degree of pain (on a scale of 0-10), number of episodes of bleeding, number of infection, and incidence of tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Tiger, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Medical Center Peabody, Peabody, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Final results will be shared with another investigator who will not be participating in the clinical trial but will author the paper. All individual participant data will be de-identified before sharing with this investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available once the final patient has finished the study and the data has been compiled and de-identified. It will be available until the paper is accepted for publication.
Access Criteria: Investigator will have access to the results as needed to author the paper.

REFERENCES:
- [Background] Saap LJ, Falanga V. Debridement performance index and its correlation with complete closure of diabetic foot ulcers. Wound Repair Regen. 2002 Nov-Dec;10(6):354-9. doi: 10.1046/j.1524-475x.2002.10603.x. PMID 12453138
- [Background] Steed DL. Debridement. Am J Surg. 2004 May;187(5A):71S-74S. doi: 10.1016/S0002-9610(03)00307-6. PMID 15147995
- [Background] Hess CT, Kirsner RS. Orchestrating wound healing: assessing and preparing the wound bed. Adv Skin Wound Care. 2003 Sep-Oct;16(5):246-57; quiz 258-9. doi: 10.1097/00129334-200309000-00015. PMID 14581817
- [Background] Fonder MA, Lazarus GS, Cowan DA, Aronson-Cook B, Kohli AR, Mamelak AJ. Treating the chronic wound: A practical approach to the care of nonhealing wounds and wound care dressings. J Am Acad Dermatol. 2008 Feb;58(2):185-206. doi: 10.1016/j.jaad.2007.08.048. PMID 18222318
- [Background] Alavi A, Sibbald RG, Phillips TJ, Miller OF, Margolis DJ, Marston W, Woo K, Romanelli M, Kirsner RS. What's new: Management of venous leg ulcers: Treating venous leg ulcers. J Am Acad Dermatol. 2016 Apr;74(4):643-64; quiz 665-6. doi: 10.1016/j.jaad.2015.03.059. PMID 26979355
- [Background] Wilcox JR, Carter MJ, Covington S. Frequency of debridements and time to heal: a retrospective cohort study of 312 744 wounds. JAMA Dermatol. 2013 Sep;149(9):1050-8. doi: 10.1001/jamadermatol.2013.4960. PMID 23884238
- [Background] Luft HS. Becoming accountable-opportunities and obstacles for ACOs. N Engl J Med. 2010 Oct 7;363(15):1389-91. doi: 10.1056/NEJMp1009380. No abstract available. PMID 20925539
- [Background] Gloster HM Jr. The use of second-intention healing for partial-thickness Mohs defects involving the vermilion and/or mucosal surfaces of the lip. J Am Acad Dermatol. 2002 Dec;47(6):893-7. doi: 10.1067/mjd.2002.125065. PMID 12451375
- [Background] Gohari S, Gambla C, Healey M, Spaulding G, Gordon KB, Swan J, Cook B, West DP, Lapiere JC. Evaluation of tissue-engineered skin (human skin substitute) and secondary intention healing in the treatment of full thickness wounds after Mohs micrographic or excisional surgery. Dermatol Surg. 2002 Dec;28(12):1107-14; discussion 1114. doi: 10.1046/j.1524-4725.2002.02130.x. PMID 12472488
- [Background] Dodson MK, Magann EF, Meeks GR. A randomized comparison of secondary closure and secondary intention in patients with superficial wound dehiscence. Obstet Gynecol. 1992 Sep;80(3 Pt 1):321-4. PMID 1495686
- [Background] Joo J, Custis T, Armstrong AW, King TH, Omlin K, Kappel ST, Eisen DB. Purse-string suture vs second intention healing: results of a randomized, blind clinical trial. JAMA Dermatol. 2015 Mar;151(3):265-70. doi: 10.1001/jamadermatol.2014.2313. PMID 25372450
- [Background] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03880331/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03880331/ICF_003.pdf